CLINICAL TRIAL: NCT04442828
Title: 3D Echocardiography and Cardiovascular PRognosis In Mitral REgurgitation (3D-PRIME)
Brief Title: 3D Echocardiography and Cardiovascular Prognosis in Mitral Regurgitation
Acronym: 3D-PRIME
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 106848
Record Dates: First submitted 2020-06-19; First posted 2020-06-23 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Proteomics, metabolomics
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary mitral regurgitation: Patients with mitral regurgitation due to mitral valve disease
  Interventions: Diagnostic Test: Use of 3D echocardiography in patient follow-up
- Secondary mitral regurgitation: Patients with mitral regurgitation due to ventricular or atrial disease
  Interventions: Diagnostic Test: Use of 3D echocardiography in patient follow-up

INTERVENTIONS:
Diagnostic Test: Use of 3D echocardiography in patient follow-up — Patients will undergo clinical and echocardiographic examination including detailed 3D echocardiography at study inclusion and at least one follow-up visit.

SUMMARY:
The 3D-PRIME study will analyse whether use of 3D echocardiography can improve risk stratification and cardiovascular outcome in patients with mitral regurgitation of different etiologies.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with primary or secondary mitral regurgitation (MR)
* MR of moderate or severe degree
* 3D echocardiographic examinations of >= good spatial and temporal resolution

Exclusion Criteria:

* Co-existence of another valve disease of severe degree
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A cohort of patients with chronic mitral regurgitation referred for clinical and echocardiographic assessment at the Heart Valve Clinic at Haukeland University Hospital in Bergen, Norway.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-04-17 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Major cardiovascular event | 24 months
  Death, mitral valve intervention, heart failure hospitalization

SECONDARY OUTCOMES:
All-cause death | 24 months
Cardiovascular death | 24 months
Mitral valve intervention | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berg-Hansen CE, Sindre RB, Grymyr LMD, Rogge B, Valeur AE, Urheim S, Hung J, Cramariuc D. Sex differences in left atrial volumes, mechanics, and stiffness in primary mitral regurgitation-a combined 2D and 3D echocardiographic study. Eur Heart J Cardiovasc Imaging. 2024 Jul 31;25(8):1118-1126. doi: 10.1093/ehjci/jeae072. PMID 38469654